CLINICAL TRIAL: NCT03075618
Title: Acute Pancreatitis Patient Registry To Examine Novel Therapies In Clinical Experiences (APPRENTICE)
Acronym: APPRENTICE
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, David Whitcomb, Professor of Medicine, University of Pittsburgh
Other Study IDs: PRO15040389
Record Dates: First submitted 2017-02-02; First posted 2017-03-09 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples will be obtained to study DNA.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Acute Pancreatitis: Patients with Acute Pancreatitis.
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — Questionnaires

SUMMARY:
The management of acute pancreatitis is mainly based on expert opinions; large randomized controlled trials are missing and novel therapeutic approaches are considered necessary. This study will evaluate the current management and outcomes of acute pancreatitis around the world.

DETAILED DESCRIPTION:
The initial study design with discussions about the different variables to be included into the investigators' prospective database started during 2014 PancreasFest held in Pittsburgh, PA in late July 2014 under the sponsorship of Collaborative Alliance for Pancreatic Education and Research (CAPER). Following this, a datasheet with variables was created, distributed through the initial participants, and further suggestions and edits were made. The investigators now plan to move ahead with a web based seminar. All previous participants, as well as new investigators/centers that have shown interest in participating throughout the world will be invited. The webinar will be chaired by Dr. Papachristou at the University of Pittsburgh and again sponsored by CAPER. The investigators plan to discuss previous experience with collaborative, multi-continent, clinical studies in pancreas research, details of IRB submission, access and technical aspects of REDCap, and review the current datasheet for any further edits needed.

Following this, each investigator will initiate the process of applying for approval to the Institutional Review Board of his/her center. University of Pittsburgh will share their accepted, ongoing PROOF protocol as a reference. Investigators/centers with active protocol approval will start enrolling patients. The investigators plan to have a Webinar every 3-4 months and/or schedule a working group meeting at DDW in May 2015 and/or EPC in June 2015 pending on attendance of these meetings by the investigators. Finally, the investigators will present all the above steps and the progress made by our working group in 2015 PancreasFest in Pittsburgh, PA.

The initial aim of this study is to develop a core of highly motivated investigators throughout the world and enroll large number of subjects into an Internet-based database. The study team plans to monitor data recording closely and prepare our first manuscript when we reach a critical number of patients. The future goal is to maintain this collaborative core and expand into designing randomized controlled trials addressing critical questions in the management of acute pancreatitis as well as applying for funding.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of AP based upon presence of two out of the three following criteria:

   1. Abdominal pain typical to AP
   2. Serum amylase or lipase levels more than three times the upper limit of normal
   3. Imaging findings suggestive of AP
2. Willingness to participate in the study and ability to sign informed consent by patient or his/her proxy (if unable to speak).

Exclusion Criteria:

1. Age under 18 years
2. Unwilling to provide consent by patient or his/her proxy
3. Presence of pancreatic cancer
4. Presence of chronic pancreatitis
5. Occurrence of AP following a multiple trauma episode
6. Having history of organ transplant
7. Presence of any cancer which required chemotherapy or radiation therapy in the past year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Acute Pancreatitis, ages 18 and over.
Sampling Method: Probability Sample
Enrollment: 623 (Actual)
Dates: Start 2015-07; Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Number of patients with persistent organ failure as assessed by their clinical course. | 12 months
  Evaluation of the existing risks, predictive scores, and markers of severe disease.
Number of patients with pancreatic necrosis as assessed by their clinical course. | 12 months
  Evaluation of the existing risks, predictive scores, and markers of severe disease.
Number of patients with persistent organ failure as assessed by their clinical course. | 12 months
  Evaluation of the current management and outcomes of acute pancreatitis around the world.
Number of patients with pancreatic necrosis as assessed by their clinical course. | 12 months
  Evaluation of the current management and outcomes of acute pancreatitis around the world.

CONTACTS AND LOCATIONS:
Overall Officials: George Papachristou, MD, Study Chair — Ohio State University
Locations (1):
- UPMC Presbyterian, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
Findings will be shared with co-collaborators and the Collaborative Alliance for Pancreatic Education and Research.

REFERENCES:
- [Derived] Lee PJ, Culp S, Kamal A, Paragomi P, Pothoulakis I, Talukdar R, Kochhar R, Goenka MK, Gulla A, Gonzales J, Stevens T, Barbu S, Nawaz H, Gutierrez S, Zarnescu N, Capurso G, Easler J, Triantafyllou K, Ocampo C, de-Madaria E, Wu B, Hart PA, Akshintala VS, Singh VK, Bischof J, Buxbaum J, Pelaez M, Papachristou GI. Lactated Ringers Use in the First 24 Hours of Hospitalization Is Associated With Improved Outcomes in 999 Patients With Acute Pancreatitis. Am J Gastroenterol. 2023 Dec 1;118(12):2258-2266. doi: 10.14309/ajg.0000000000002391. Epub 2023 Jul 10. PMID 37428139
- [Derived] Paragomi P, Tuft M, Pothoulakis I, Singh VK, Stevens T, Nawaz H, Easler JJ, Thakkar S, Cote GA, Lee PJ, Akshintala V, Kamal A, Gougol A, Phillips AE, Machicado JD, Whitcomb DC, Greer PJ, Buxbaum JL, Hart P, Conwell D, Tang G, Wu BU, Papachristou GI. Dynamic changes in the pancreatitis activity scoring system during hospital course in a multicenter, prospective cohort. J Gastroenterol Hepatol. 2021 Sep;36(9):2416-2423. doi: 10.1111/jgh.15430. Epub 2021 Feb 18. PMID 33604947
- [Derived] Matta B, Gougol A, Gao X, Reddy N, Talukdar R, Kochhar R, Goenka MK, Gulla A, Gonzalez JA, Singh VK, Ferreira M, Stevens T, Barbu ST, Nawaz H, Gutierrez SC, Zarnescu NO, Capurso G, Easler J, Triantafyllou K, Pelaez-Luna M, Thakkar S, Ocampo C, de-Madaria E, Cote GA, Wu BU, Paragomi P, Pothoulakis I, Tang G, Papachristou GI. Worldwide Variations in Demographics, Management, and Outcomes of Acute Pancreatitis. Clin Gastroenterol Hepatol. 2020 Jun;18(7):1567-1575.e2. doi: 10.1016/j.cgh.2019.11.017. Epub 2019 Nov 9. PMID 31712075